CLINICAL TRIAL: NCT02105402
Title: Treatment Efficacy for Developmental Motor Speech Disorders: A PROMPT Randomized Control Trial
Brief Title: Treatment Efficacy for Developmental Motor Speech Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Prompt Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROMPT-29142
Record Dates: First submitted 2014-04-01; First posted 2014-04-07 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Randomized Controlled Trial for Speech Disorders in Children
Keywords: Speech sound disorders; Randomized Controlled Trial; Speech intelligibility; PROMPT treatment; Developmental motor speech disorders; Children; Functional outcomes; Treatment efficacy
MeSH Terms: conditions — Speech Sound Disorder; Speech Intelligibility

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group - PROMPT therapy (Experimental): Prompts for Restructuring Oral Muscular Phonetic Targets (PROMPT)
  Interventions: Behavioral: PROMPT
- Waitlist or Delay Group (No Intervention): Participants in this group are on the waitlist for 10 weeks

INTERVENTIONS:
Behavioral: PROMPT — The PROMPT approach utilizes a motor-speech hierarchy (MSH) to guide speech language pathologists (SLP) in selecting speech movement goals for treatment. PROMPT treatment generally proceeds systematically in a bottom-up fashion starting with the lowest subsystem in the hierarchy where a child has control issues. Furthermore, in the PROMPT approach specific techniques are used to stimulate sensory input that are assumed to facilitate the formation of sensory-motor pathways required for the acquisition and accurate production of speech movement patterns. As the speech motor behaviors are established, the clinician reduces the number of cues and the frequency and immediacy of feedback and practices transfer and generalization activities.
  Other Names: PROMPT therapy
  Arms: Intervention Group - PROMPT therapy

SUMMARY:
The purpose of this study is to carry out a high-level treatment efficacy study on children with speech sound disorders with motor speech involvement (SSD-MSI) using a well-controlled Randomized Controlled Trial design.

The intervention of choice is the Prompts for Restructuring Oral Muscular Phonetic Targets (PROMPT) approach, which has been effective in treating motor speech disorders in adults and in children with autism and cerebral palsy.

DETAILED DESCRIPTION:
The results of this study will allow us to determine if there is a causal relationship between PROMPT treatment and outcome measures and predict how much improvement can be expected from this therapy. This study is being conducted as a part of a multicenter clinical trial in the province of Ontario, Canada with three sites: The John McGivney Children's Centre in Windsor, The ErinoakKids Centre for Treatment and Development in Mississauga, and The Speech and Stuttering Institute in Toronto.

The study integrity will be monitored by an arms-length, external agency, The Applied Health Research Centre (AHRC) at St. Michael's Hospital in Toronto. The study is coordinated by the Department of Speech-Language Pathology at the University of Toronto and funded by the PROMPT Institute in Santa Fe, New Mexico.

ELIGIBILITY:
Inclusion Criteria:

* The child is between 3 and 10 Years.
* English is the primary language spoken by the primary caregiver at home.
* Hearing/Vision (corrected is acceptable- e.g., spectacles) is within normal limits.
* Readiness for direct speech therapy.
* Age appropriate social interaction and play skills.
* Age appropriate or mildly delayed receptive language skills.
* Normal to any amount of delay in expressive language development.
* Moderate to severe speech sound disorder.
* Age appropriate or slight delay non-verbal intelligence.
* 4 red flags for motor speech involvement.

Exclusion Criteria:

* Signs and symptoms suggesting global motor involvement (Cerebral Palsy).
* Signs and symptoms suggesting Autism Spectrum Disorders.
* Oral structural deficits.
* Feeding impairments.
* Signs of Dysarthric speech or significant drooling.
* Prosodic and / or resonance disorders.
* Diagnosis of Childhood Apraxia of Speech features

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in speech motor control | At baseline and following 10 weeks of intervention or waitlist delay
  Formal assessment of the neuromotor integrity of the motor speech system will be carried out using the verbal motor production assessment for children (VMPAC).
Change in speech articulation | At baseline and following 10 weeks of intervention or waitlist delay
  Assessment of speech articulation will be carried out using the Diagnostic Evaluation of Articulation and Phonology (DEAP) test.
Change in word-level speech intelligibility | At baseline and following 10 weeks of intervention or waitlist delay
  Word level assessment of speech intelligibility will be carried out using the Children's speech Intelligibility Measure.
Change in Functional Communication: | At baseline and following 10 weeks of intervention or waitlist delay
  Focus on the Outcomes of Communication Under Six (FOCUS), is a parent questionnaire that captures preschool children's communication abilities as they participate in real-world situations.
Change in criterion-referenced measure of speech motor control. | At baseline and following 10 weeks of intervention or waitlist delay
  Criterion-referenced assessment of the motor speech system will be carried out using a set of probe words. The audio-video recordings of the probe words will be analyzed by three qualified and blinded speech language pathologists.
Change in phonological processes | At baseline and following 10 weeks of intervention or waitlist delay
  Phonological processes will be assessed using the Diagnostic Evaluation of Articulation and Phonology (DEAP) test.
Change in sentence-level speech intelligibility | At baseline and following 10 weeks of intervention or waitlist delay
  Sentence-level assessment of speech intelligibility will be carried out using the Beginner's Intelligibility Test.

CONTACTS AND LOCATIONS:
Overall Officials: Aravind Namasivayam, Ph.D., Principal Investigator — University of Toronto; Deborah Hayden, M.A., Study Director — The PROMPT Institute, Santa Fe, NM, 87505 USA; Pascal van Lieshout, Ph.D., Study Chair — University of Toronto
Locations (3):
- Canada (3):
  - ErinoakKids Centre for Treatment and Development, Mississauga, Ontario
  - The Speech and Stuttering Institute, Toronto, Ontario
  - The John McGivney Children's Centre of Essex County, Windsor, Ontario